CLINICAL TRIAL: NCT05546632
Title: Evaluation of Cyto-chex Tubes for the Measurement of Monocyte Expression of HLA-DR Molecules by Flow Cytometry
Brief Title: Evaluation of Cyto-chex Tubes for the Measurement of Monocyte Expression of Human Leukocyte Antigen - DR Isotype (HLA-DR) Molecules by Flow Cytometry
Acronym: CHEX-DR
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0446
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Critical Care
Keywords: Intensive care unit; HLA-DR; blood sample; Cyto-chex tube; EDTA tube
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill patients: Patients included in this study will have blood sampling using EDTA tube and nex generation Cyto-Chex BCT tubes in order to compare compare the expression of mHLA-DR with these two types of tubes
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — Patients will have one blood sampling using one EDTA tube and one Cyto-Chex BCT tube, one after the other

SUMMARY:
The expression of mHLA-DR, measured by flow cytometry, is today the reference marker to guide immunostimulatory therapies (IFN-γ) in the most severely immunocompromised patients. Nevertheless, pre-analytical constraints (storage of samples at +4°C before analysis) limit the wide use of mHLA-DR in clinical practice (problem of transporting samples to sites with a flow cytometer). Recent studies have shown that samples taken on Cyto-Chex Blood Collection Tubes (BCT) (containing a cell membrane stabilizer) were, for mHLA-DR, stable at room temperature during 72 hours after sampling. The main objective of this study is to compare the expression of mHLA-DR from samples taken simultaneously from standard tubes (EDTA) and new generation Cyto-Chex BCT tubes, to validate using Cyto Chex BCT tube in the clinical practice.

The investigators think that mHLA-DR quantification performed from Cyto-Chex BCT tubes is reliable and similar to quantification performed from EDTA tubes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient hospitalized in intensive care unit
* Patient able to consent and having expressed his non-objection (in the case where the patient is aware) OR Patient whose trusted person has given his non-objection (in the case where the patient is not able to consent, example intubated patient)

Exclusion Criteria:

* Pregnant women
* Minors
* Persons deprived of their liberty by a judicial or administrative decision
* Persons subject to psychiatric care
* Adults subject to a legal protection measure (guardianship, protection of vulnerable adults)
* Patient who doesn't understand French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will focus on patients hospitalized in the intensive care unit of the Edouard Herriot hospital in Lyon
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Quantity of anti-HLA-DR antibodies per cell | The day of inclusion
  The quantity of anti-HLA-DR antibodies per single cell will be assessed in each tube (EDTA and Cyto Chex) using flowcytometry

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Claire LUKASZEWICZ, Professor, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service de reanimation chirurgicale, Lyon, France

IPD SHARING:
Plan to Share IPD: No